CLINICAL TRIAL: NCT05444335
Title: Screening for Atrial Fibrillation in Elderly Women Older Than 70 Years
Acronym: SAFE-W
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Prachi Mehndiratta, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HP-00099005
Record Dates: First submitted 2022-06-22; First posted 2022-07-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation New Onset

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention arm (Other): Women older than 70 who would wear the Zio patch for 2 weeks
  Interventions: Device: Wearable cardiac monitor -Zio patch

INTERVENTIONS:
Device: Wearable cardiac monitor -Zio patch — Women older than 70 years old will be asked to wear a cutaneous cardiac monitor for 2 weeks.

SUMMARY:
Screening for Atrial Fibrillation in Elderly Women (SAFE-W) is a pilot study evaluating the prevalence of atrial fibrillation (Afib) in a rapidly aging segment of the population. Studies have shown that women with Afib are more likely to be symptomatic, have increased mortality from stroke resulting from Afib, and are less likely to receive treatment for Afib. University of Maryland Department of Neurology and Vascular Neurology are recruiting women older than 70 years of age to participate in the study.

DETAILED DESCRIPTION:
Atrial fibrillation or irregular heart beat is seen in 1/3rd of patients that present with stroke. Atrial fibrillation is being increasingly seen in women older than 70 as women are likely to live longer. Women are more likely to die from atrial fibrillation related stroke and are more likely to have symptoms from uncontrolled atrial fibrillation. They are also less likely to be treated with blood thinners to prevent stroke. This section of the population has been underrepresented in other studies on atrial fibrillation and the aim of this study is to proactively screen women older than 70 who are at risk for atrial fibrillation by using a wearable cardiac monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Female sex
2. No previous diagnosis of atrial fibrillation
3. Age ≥70 years
4. CHA2DS2-VASc score ≥4

Exclusion Criteria:

1. Life expectancy < 2 years
2. Dementia or other neurologic condition which would make outpatient follow-up difficult
3. CHA2DS2-VASc score ≤3
4. Any compliance issues - such as heavy alcohol/drug use that would impede follow up.

Ages: 70 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Women
Enrollment: 120 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Rate of detection of atrial fibrillation | 1 year
  Percentage of women older than 70 found to have atrial fibrillation one year from enrollment
Anticoagulant use for prevention of stroke | 2 years
  Rate of anticoagulant prescription

SECONDARY OUTCOMES:
Device adherence | 1 year
  Rate of compliance with device - participants would be asked if they wore the device as advised for the two weeks and adherence would be reported as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Prachi Mehndiratta, MBBS, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrade JG, Deyell MW, Lee AYK, Macle L. Sex Differences in Atrial Fibrillation. Can J Cardiol. 2018 Apr;34(4):429-436. doi: 10.1016/j.cjca.2017.11.022. Epub 2017 Dec 6. PMID 29455950
- [Background] Madsen TE, Howard VJ, Jimenez M, Rexrode KM, Acelajado MC, Kleindorfer D, Chaturvedi S. Impact of Conventional Stroke Risk Factors on Stroke in Women: An Update. Stroke. 2018 Mar;49(3):536-542. doi: 10.1161/STROKEAHA.117.018418. Epub 2018 Feb 8. No abstract available. PMID 29438086
- [Background] Gladstone DJ, Wachter R, Schmalstieg-Bahr K, Quinn FR, Hummers E, Ivers N, Marsden T, Thornton A, Djuric A, Suerbaum J, von Grunhagen D, McIntyre WF, Benz AP, Wong JA, Merali F, Henein S, Nichol C, Connolly SJ, Healey JS; SCREEN-AF Investigators and Coordinators. Screening for Atrial Fibrillation in the Older Population: A Randomized Clinical Trial. JAMA Cardiol. 2021 May 1;6(5):558-567. doi: 10.1001/jamacardio.2021.0038. PMID 33625468